CLINICAL TRIAL: NCT06938997
Title: The Effectiveness of Combining AR/VR Technology in Virtual Clinical Auditory Hallucinations on the Comprehensive Auditory Hallucination Nursing Competency of Psychiatric Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: NYCU113052AE
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Nurses; Schizophenia Disorder; Hallucinations, Auditory
Keywords: Auditory hallucination care competence; virtual reality; schizophrenia; Objective Structured Clinical Examination
MeSH Terms: conditions — Hallucinations; Schizophrenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50-minute Auditory Hallucination Care instructional video (Placebo Comparator): Control Group
  * Pre-test: No intervention
  * Intervention 1: Auditory Hallucination Care Video only
  * Post-test: Conduct measurement (no new intervention)
  * Intervention 2: 50-minute Auditory Hallucination Care instructional video only
  * Follow-up: Conduct measurements (no new intervention)
  Interventions: Other: Auditory Hallucination Care Video
- Virtual clinical auditory hallucination solution and Auditory Hallucination Care instructional vide (Experimental): Experimental Group
  * Pre-test: No intervention
  * Intervention 1: Accept intervention A+B
  * A: Virtual clinical auditory hallucination solution combining AR/VR technology and virtual human interactive platform
  * B: 50-minute Auditory Hallucination Care instructional video
  * Post-test: Conduct measurement (no new intervention)
  * Intervention 2: Re-intervention of A+B
  * Follow-up: Conduct measurements (no new intervention)
  Interventions: Other: Virtual clinical auditory hallucination solution combining AR/VR technology; Other: Auditory Hallucination Care Video

INTERVENTIONS:
Other: Virtual clinical auditory hallucination solution combining AR/VR technology — This study, titled "Effectiveness of AR/VR-integrated OSCE on Psychiatric Nurses' Comprehensive Auditory Hallucination Care Ability: A Randomized Controlled Trial," involves both experimental and control groups watching videos. The control group views standard educational videos, while the experimental group uses AR/VR technology, virtual patient interaction platforms, and educational videos in a simulated clinical environment. Four scripts were developed: two for training and two for pre/post-testing. All scripts and OSCE checklists are researcher-developed, reviewed by experts, and pilot tested.
  Arms: Virtual clinical auditory hallucination solution and Auditory Hallucination Care instructional vide
Other: Auditory Hallucination Care Video — The videos include professional knowledge and skills related to auditory hallucinations.

SUMMARY:
This study aims to develop and evaluate a Virtual Reality (VR) Auditory Hallucination Program to enhance psychiatric nurses' comprehensive care competence in managing auditory hallucinations among patients with schizophrenia. Given that 60-80% of patients on the schizophrenia spectrum experience auditory hallucinations, and many continue to do so despite medication, improving nurses' professional skills in this area is critical.

The research is conducted in two phases across four psychiatric institutions. Phase one involves the development and validation of the VR program and an OSCE (Objective Structured Clinical Examination), piloted with five participants and evaluated by psychiatric nursing experts. Phase two is a formal interventional study with 200 psychiatric nurses, using block randomization and three data collection time points.

Assessment tools include five instruments measuring nurses' confidence, knowledge, attitude, empathy, immersion, and care performance related to auditory hallucinations. The study expects to strengthen nurses' ability to assess and manage auditory hallucinations effectively, and proposes the VR program as a potential tool for nursing in-service education.

DETAILED DESCRIPTION:
Background: The lifetime prevalence of auditory hallucinations among patients on the schizophrenia spectrum is 60-80%. More than half of these patients continue to experience auditory hallucinations even with regular medication adherence. The professional competence of nurses in managing auditory hallucinations affects the stability of patients' symptoms and their recovery process, highlighting the importance of nurses' capabilities in caring for patients with auditory hallucinations.

Purpose: To develop and test the effectiveness of a virtual reality auditory hallucination program on the comprehensive care competence of psychiatric nurses in managing auditory hallucinations.

Methods: This is a two-phase study conducted in four psychiatric medical institutions. The study includes a development phase, a testing phase, and a formal research phase. In the pilot phase, five participants are expected to be recruited. The first phase involves the development and testing of the virtual reality auditory hallucination program and the Objective Structured Clinical Examination (OSCE), which includes components such as auditory hallucination assessment, communication with individuals experiencing auditory hallucinations, and management of auditory hallucinations. Upon completion, content validation will be conducted by psychiatric experts. Five psychiatric nursing master's students will be invited as simulated candidates to examine the applicability of the "VR-based Auditory Hallucination Nursing OSCE" for psychiatric nurses. The second phase is the formal interventional study, which will recruit 200 psychiatric nurses through convenience sampling. Participants will be grouped by institution using block randomization software. Data will be collected at three time points using the HTC virtual human system in conjunction with Google online questionnaires. The research instruments include:

* Self-rated Confidence Questionnaire on Auditory Hallucination Assessment and Management,② Auditory Hallucination Knowledge, Attitude, and Empathy Self-awareness Scale,③ Auditory Hallucination Immersion and Empathy Scale, ④ Comprehensive Auditory Hallucination Nursing OSCE Evaluation Form, and ⑤ Nurse Auditory Hallucination Literacy Scale. Expected Results: This study is expected to enhance psychiatric nurses' capabilities in assessing and managing auditory hallucinations. The program may be routinely used in in-service education for nursing staff and may serve as a reference to assist nurses in helping patients improve their insight into auditory hallucinations.

Keywords: Auditory hallucination care competence, interventional study, virtual reality, schizophrenia, Objective Structured Clinical Examination (OSCE)

ELIGIBILITY:
Inclusion Criteria:

* A psychiatric nurse who has been engaged in nursing work in a psychiatric unit for at least three months;
* Those who were willing to participate in the study and filled out the consent form;
* Willing to use smartphones to watch VR360 videos;
* Willing to cooperate with the study and use 3D glasses.

Exclusion Criteria:

* Nurses who are about to leave or be transferred out of the psychiatric ward within six months
* Part-time nurses
* Part-time supervisors
* Specialist nurses.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Auditory Hallucination Immersion and Empathy Scale | At baseline (pre-intervention), 6 weeks after the first intervention, and 6 weeks after the second intervention.
  To assess the impact of the intervention on empathy, this study uses the Situational Scale of Empathetic Responses (Schutte & Stilinović, 2017), consisting of 15 items-7 on empathic perspective taking and 8 on empathic concern. Participants imagine interacting with a person hearing voices and rate items on a 5-point Likert scale (1 = strongly disagree to 5 = strongly agree); higher scores indicate greater empathy in auditory hallucination scenarios. The scale was translated and validated for content. Additionally, we will adopt the Jefferson Scale of Empathy (JSE-HP version), translated and adapted by Cheng et al. (2011), with a KMO of 0.93 and Cronbach's α = .73-.89.
Auditory Hallucination Knowledge, Attitude, and Empathic Self-Awareness Scale; Auditory Hallucination Literacy Scale. | At baseline (pre-intervention), 6 weeks after the first intervention, and 6 weeks after the second intervention.
  This tool, developed by Mawson (2014), includes 11 items assessing knowledge, attitudes, and empathy toward auditory hallucinations. Participants respond using a 5-point Likert scale ranging from "strongly agree" (5) to "strongly disagree" (1). As it has not been used in Taiwan, we have completed forward and backward translation and content validity testing. Reliability and validity testing of the Chinese version will be completed before the intervention study.

SECONDARY OUTCOMES:
Demographic variables | Before intervention
  Includes age, educational level, gender, marital status, total years of nursing experience, years of psychiatric nursing experience, advanced certifications (nurse practitioner, psychiatric mental health nurse, community psychiatric mental health nurse), level of competency advancement, workplace setting, and type of employment.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Yuli Hospital, Ministry of Health and Welfare, Hualien City
  - Tsaotun Psychiatric Center, Ministry of Health and Welfare, Nantou County
  - Bali Psychiatric Center, Ministry of Health and Welfare, New Taipei City
  - Tri-Service General Hospital Beitou Branch, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dutta TK, Veeresh A, Mathur C, Phani V, Mandal A, Sagar D, Nebapure SM. The induced knockdown of GmCAD receptor protein encoding gene in Galleria mellonella decreased the insect susceptibility to a Photorhabdus akhurstii oral toxin. Virulence. 2021 Dec;12(1):2957-2971. doi: 10.1080/21505594.2021.2006996. PMID 34882066
- [Result] Lee JH, An CH, Yoo NJ, Lee SH. Mutational intratumoral heterogeneity of a putative tumor suppressor gene RARRES3 in colorectal cancers. Pathol Res Pract. 2018 Apr;214(4):601-602. doi: 10.1016/j.prp.2017.12.011. Epub 2017 Dec 21. No abstract available. PMID 29496306
- [Result] Della Libera C, Goosse M, Laroi F, Willems S. Examining the impact of experiencing auditory verbal hallucinations from a first-person perspective on the degree of empathy and stigmatization in a group of psychology students: A study using 360 degrees immersive videos. Compr Psychiatry. 2023 May;123:152379. doi: 10.1016/j.comppsych.2023.152379. Epub 2023 Feb 26. PMID 36870090
- [Result] de Leede-Smith S, Barkus E. A comprehensive review of auditory verbal hallucinations: lifetime prevalence, correlates and mechanisms in healthy and clinical individuals. Front Hum Neurosci. 2013 Jul 16;7:367. doi: 10.3389/fnhum.2013.00367. eCollection 2013. PMID 23882203
- [Result] Craig TK, Rus-Calafell M, Ward T, Leff JP, Huckvale M, Howarth E, Emsley R, Garety PA. AVATAR therapy for auditory verbal hallucinations in people with psychosis: a single-blind, randomised controlled trial. Lancet Psychiatry. 2018 Jan;5(1):31-40. doi: 10.1016/S2215-0366(17)30427-3. Epub 2017 Nov 23. PMID 29175276
- [Result] Carlson CG. Virtual and Augmented Simulations in Mental Health. Curr Psychiatry Rep. 2023 Sep;25(9):365-371. doi: 10.1007/s11920-023-01438-4. Epub 2023 Aug 25. PMID 37624512
- [Result] Browne C, Wall P, Walters J. Exploring Nursing Students' Experiences With Different Teaching Pedagogies: A Mixed-Methods Study. J Nurs Educ. 2022 Mar;61(3):147-152. doi: 10.3928/01484834-20220109-04. Epub 2022 Mar 1. PMID 35254159
- [Result] Abdolrahimi M, Ghiyasvandian S, Zakerimoghadam M, Ebadi A. Therapeutic communication in nursing students: A Walker & Avant concept analysis. Electron Physician. 2017 Aug 25;9(8):4968-4977. doi: 10.19082/4968. eCollection 2017 Aug. PMID 28979730